CLINICAL TRIAL: NCT01946035
Title: A Proof of Concept Study in Allergic Rhinitis, to Evaluate the Differential Effects Between Single and Chronic Dosing of Doxazosin on Nasal Airway Calibre
Brief Title: Alpha-Blockers in Allergic Rhinitis (MAN 01)
Acronym: MAN01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, Brian J Lipworth, Professor of Allergy and Pulmonology, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012RC14
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will take 1 capsule placebo each evening
  Interventions: Other: Placebo
- Doxazosin XL (Experimental): Participants will take 1 capsule Doxazosin 4mg XL each evening
  Interventions: Drug: Doxazosin XL

INTERVENTIONS:
Drug: Doxazosin XL
  Other Names: Cardozin XL 4mg Prolonged-release Tablets
  Arms: Doxazosin XL
Other: Placebo
  Arms: Placebo

SUMMARY:
Allergic rhinitis (allergic inflammation of the nose) is a common medical condition which is known to seriously decrease quality of life, aggravate preexisting conditions particularly asthma, carry significant medical treatment costs and be responsible for reduced work productivity and lost school days. A significant symptom of the condition, nasal blockage, remains difficult to treat even when using nasal corticosteroids. Decongestant medications act on the blood vessels in the nose and have an immediate effect in clearing a blocked nose but if used for more than seven days a more severe rebound congestion of the nose develops.

In this study, the investigators aim to assess the effects of doxazosin, a drug which is currently used to treat high blood pressure and symptoms of prostate enlargement, to find out if it has an effect on nasal blockage.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-70 years
* Able to provide informed consent
* Able to comply with the requirements of the protocol
* Diagnosis of allergic rhinitis
* Peak nasal inspiratory flow which is reversible to >20 l/min with oxymetazoline
* Positive skin prick test to at least one common aeroallergen
* Ability to withhold antihistamines, intranasal corticosteroids for duration of the study
* Agreement for their GP to be made aware of study participation and to receive feedback as relevant to the participant's well being

Exclusion Criteria:

* Pregnancy, planned pregnancy or lactation
* Respiratory tract infection in the previous 2 months
* Nasal polyps of more than Grade I on nasal endoscopy
* Any known adverse reaction to the Investigational Medicinal Product or other quinazolines
* Systolic BP <100mmHg
* Any degree of heart block
* Any clinically significant medical condition that may endanger the health or safety of the participant or jeopardise the protocol
* Participation within another clinical trial of investigational medicinal product within the last 30 days
* Under the age of 18
* Benign hyperplasia, chronic urinary tract infections, bladder stones, overflow bladder, anuria or progressive renal failure
* History of oesophageal or gastrointestinal obstruction or decreased lumen diameter of the gastrointestinal tract.
* Concomitant use of PDE5 inhibitors (sildenafil etc.)
* Alpha antagonists - this is the medication under investigation.
* Other cardiovascular medications including but not limited to:

ACE inhibitors, Angiotensin II antagonists, Beta blockers, calcium channel blockers, diuretics, nitrates, phosphodiesterase type-5 inhibitors or other vasodilating medications - these in combination with doxazosin carry an increased risk of symptomatic hypotension.

* Monoamine oxidase inhibitors (MAOIs) - antidepressant medication that can lead to significant hypotension in combination with alpha antagonists.
* Anxiolytics and hypnotics - enhanced hypotensive and sedative effects when alpha-blockers given in combination with these.
* Methyldopa and levodopa - potential enhanced hypotensive effect with alpha antagonists.
* Nasal corticosteroid spray - would confound study outcomes
* Oxymetazoline - this is used as an outcome of response in the study.
* Antihistamines - the participants will be undergoing a histamine nasal challenge.
* Sympathomimetics i.e. dopamine, ephedrine, epinephrine, metaraminol, methoxamine, phenylephrine- may reduce the effect of doxazosin.
* Any other medication, which in the opinion of the Investigator may put the participant at risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in peak nasal inspiratory from baseline as compared with acute and chronic dosing of doxazosin versus placebo | 12 hours; 3 to 5 weeks

SECONDARY OUTCOMES:
Nasal histamine challenge response as measured by peak nasal inspiratory flow after chronic dosing | 12 hours; 3 to 5 weeks
Nasal airways resistance after single and chronic dosing | 12 hours; 3 to 5 weeks
Domiciliary peak nasal inspiratory measurements after chronic dosing | 12 hours; 3 to 5 weeks
Symptoms after chronic dosing | 12 hours; 3 to 5 weeks
Mini Rhinoconjunctivitis Quality of Life Questionnaire after chronic dosing | 24 hours; 3 to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Lipworth, MD, Principal Investigator — University of Dundee; Arvind Manoharan, MBChB, Principal Investigator — University of Dundee
Locations (1):
- Brian Lipworth, Dundee, United Kingdom

REFERENCES:
- [Background] Manoharan A, Morrison AE, Lipworth BJ. Effects of the inverse alpha-agonist doxazosin in allergic rhinitis. Clin Exp Allergy. 2016 May;46(5):696-704. doi: 10.1111/cea.12700. PMID 26741127